CLINICAL TRIAL: NCT01530464
Title: The Safety Evaluation of Aminophylline and Ambrisentan When Administered Orally Alone and in Combination to Healthy Volunteers
Acronym: GQ01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thies Schroeder (Other)
Responsible Party: Sponsor-Investigator, Thies Schroeder, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00028417
Record Dates: First submitted 2012-02-01; First posted 2012-02-10 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-11

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: High altitude induced fatigue; High altitude induced pulmonary Hypertension
MeSH Terms: conditions — Pulmonary edema of mountaineers | interventions — Aminophylline; ambrisentan

ARMS (3):
- Aminophylline (Active Comparator)
  Interventions: Drug: Aminophylline
- Ambrisentan (Active Comparator)
  Interventions: Drug: Ambrisentan
- Aminophylline and ambrisentan (Experimental): Treatment 3: Aminophylline, 500 mg plus Ambrisentan, 5 mg
  Interventions: Drug: Aminophylline plus ambrisentan

INTERVENTIONS:
Drug: Aminophylline — Drug will be administered as a single oral dose of 500mg, followed by a 48h washout period.
  Arms: Aminophylline
Drug: Ambrisentan — Drug will be administered as a single dose of 5mg, followed by a 48h washout period
  Other Names: Letairis
  Arms: Ambrisentan
Drug: Aminophylline plus ambrisentan — Drugs will be given as single doses of 500mg (aminophylline) and 5mg (ambrisentan), followed by a 48h washout period
  Arms: Aminophylline and ambrisentan

SUMMARY:
This is a Phase I, three period, two sequence, open-label, randomized, crossover study, with the primary objective of testing the safety and tolerability of combined oral doses of aminophylline and ambrisentan in healthy human subjects. The secondary objective is to assess the pharmacokinetic profiles of theophylline (aminophylline) and ambrisentan when administered alone or in combination. It is hypothesized that the combination of these drugs is generally safe, and that no drug interaction can be observed.

DETAILED DESCRIPTION:
This is a Phase I, three period, two sequence, single-center, open-label, randomized, crossover study design. Periods I and II consist of the oral administration of either a single dose of aminophylline or ambrisentan alone, followed by a 48 hour wash out interval. Subsequently, Period III consists of the simultaneous administration of both drugs. All subjects are to be confined to the Duke Clinical Research Unit throughout all treatment periods [Study Day -1 to Study Day 6 (discharge)]. A sufficient number of healthy adult subjects will be consented in order to enroll 24 and complete 16 subjects who complete all three periods. Replacement of subjects is permitted, if necessary.

Qualified subjects will be randomized into one of two sequences consisting of three Periods as indicated below:

-------------Period 1-----Period 2-----Period 3

Sequence A: Treatment 1 Treatment 2 Treatment 3

Sequence B: Treatment 2 Treatment 1 Treatment 3

TREATMENTS:

Treatment 1: Aminophylline 500 mg (corresponding to 395 mg theophylline).

Treatment 2: Ambrisentan 5 mg.

Treatment 3: Aminophylline, 500 mg plus Ambrisentan, 5 mg.

After completion of each treatment period, the subjects will proceed to the next period provided no Stopping Rules criteria have been met

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent to participation in the study prior to screening. Consent will be documented by the subject's dated signature that will be counter-signed and dated by a witness. The appropriate HIPAA authorization forms must be signed and dated by the subject.
* Subjects must be healthy non-smoking adult male and female volunteers between the ages of 18 and 40 years, with a BMI of 18-30 kg/m2 and weighing at least 150 lbs. Subjects health status will be determined by the medical history, physical examination, vital signs, electrocardiogram, blood chemistry, hematology, and urinalysis performed at screening.
* Subjects must be willing to fast a minimum of 8 hours prior to screening.
* Subjects must be willing to abstain from alcohol and xanthine-containing food and beverages from the time of admission to the clinical research inpatient unit through at least 48 hours following discharge.
* Subjects must be willing to remain in the clinical research unit continuously for the inpatient portion of the study from admission to discharge.
* Women who are of non-childbearing potential, must be either surgically sterile (removal of both ovaries and/ or uterus at least 12 months prior to dosing), or naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1, with an FSH level at screening of ≥ 40 mIU/mL.
* Women of child-bearing potential must have a negative serum pregnancy test within 48 hours of receiving study drug and must agree to avoid pregnancy during study and for one month after the last dose of study drug
* Male subjects of child-fathering potential must agree to avoid causing pregnancy during study and for three months after the last dose of study drug.
* Subjects must agree not to donate blood, plasma, platelets, or any other blood components during the study and for 4 weeks after the last dose.
* Male subjects must agree not to donate sperm during the study and for 12 weeks after the last dose.

Exclusion Criteria:

* Subjects with laboratory results outside the normal range, if considered clinically significant by the Investigator. In addition, subjects must have a normal hematocrit and hemoglobin concentration and be ≥ 36% and ≥ 12.0 g/dL, respectively.
* A mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the side effects of the study drug.
* Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years.
* Unwillingness or lack of ability to comply with the protocol, or to reside in the inpatient unit during the required time period, or to cooperate fully with the Principle Investigator and site personnel.
* Use of any of the following: Any concomitant medication including oral contraceptive hormones. Subjects who have received any prescribed or non-prescribed (over-the-counter [OTC]) systemic medication, topical medications, or herbal supplements within 14 days from Day 1. St. John's Wort (hypericin) must not have been taken for at least 30 days prior to Period 1, Day 1. Any drugs, foods or substances known to be strong inhibitors or strong inducers of CYP enzymes (also known as cytochrome P450 enzymes); especially CYP 1A2, or Pgp within 30 days prior to Period 1, Day 1
* Clinically significant ECG abnormality in the opinion of the Investigator. Vital signs or clinically significant laboratory values at the screening visit that in the opinion of the Investigator would make the subject an inappropriate candidate for the study.
* Has taken any other investigational drug during the 30 days prior to the screening visit or is currently participating in another investigational clinical trial.
* Made any significant donation (including plasma) or have had a significant loss of blood within 30 or 90 days prior to Period 1, Day 1.
* History or manifestation of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematologic or other medical disorders.
* Subjects who are carriers of the Hepatitis B surface antigen (HbsAg), Hepatitis C antibody, or HIV antibody
* Serious mental or physical illness within the past year.
* Male subjects who consume more than 28 units of alcohol per week and female subjects who consume more than 21 units of alcohol per week (one unit of alcohol equals 250 mL of beer, 100 mL or a medium glass of wine, or 25 mL of spirits) or those subjects who have a significant history of alcoholism or drug/ chemical abuse within the last 2 years
* Failure to agree to abstain from alcohol, cola, tea, coffee, chocolate and other caffeinated drink/ food from 2 days before dosing and throughout confinement
* Positive results on screening tests for drugs of abuse, cotinine or alcohol at screening or the pre-dose assessment at check-in
* Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 12 months prior to Period 1, Day 1
* Women of childbearing potential who are pregnant (as based on test results) or are breast feeding
* Subjects who have a history of hypersensitivity or idiosyncratic reaction to any of the products administered during the study.
* Subjects who, in the opinion of the Investigator, should not participate in the study.
* Subjects who are employed by the DCRU
* Subjects who have a history of unexplained syncope; i.e., autonomic dysfunction.
* Subjects who have a history of hypotension, including orthostatic hypotension
* A positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody at screening.
* Lack of ability to understand verbal and/ or written English
* History of severe hypersensitivity or allergic reaction to study medication
* Failure to agree to abstain from grapefruit and grapefruit juice as well as oranges and orange juice from 10 days before the first dose and throughout the study
* History of clinically significant illness within 4 weeks prior to Day 1
* Receipt of a transfusion or any blood products within 90 days prior to Period 1, Day 1
* History of participation in another investigational study or who have participated in an investigational study within the past 30 days prior to Period 1, Day 1

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noveck, MD, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on August 1, 2011, was stopped again after delays in acquiring study drug (ambrisentan), and commenced again on February 6, 2012, until April 14, 2012.
  The study was conducted in the Duke Clinical Research Unit (DCRU).
Pre-assignment Details: The study was initiated on August 1, 2011 and stopped on August 9, 2011 after a delay in acquiring the study drug ambrisentan. None of the 24 screened subjects were randomized in this period. The trial was re-started on February 6, 2012 and completed on April 14, 2012 with the last subject being evaluated on April 30, 2012.
Groups:
- Sequence A: Period 1: First intervention (Aminophylline 500mg, 24h) Period 2: Washout (24 hours) Period 3: Second intervention (Ambrisentan 5mg, 24h) Period 4: Washout (24h) Period 5: Third intervention (Aminophylline 500mg plus ambrisentan 5mg, 24h) Period 6: Washout (24h)
- Sequence B: Period 1: First intervention (Ambrisentan 5mg, 24h) Period 2: Washout (24 hours) Period 3: Second intervention (Aminophylline 500mg, 24h) Period 4: Washout (24h) Period 5: Third intervention (Aminophylline 500mg plus ambrisentan 5mg, 24h) Period 6: Washout (24h)
Period: First Intervention (24h)
Arm/Group | Sequence A | Sequence B
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Washout (24h)
Arm/Group | Sequence A | Sequence B
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Second Intervention (24h)
Arm/Group | Sequence A | Sequence B
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Washout (24h)
Arm/Group | Sequence A | Sequence B
Started | 10 | 8
Completed | 9 (1 subject withdrew consent and left due to family emergencies) | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Third Intervention (24h)
Arm/Group | Sequence A | Sequence B
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Washout (24h)
Arm/Group | Sequence A | Sequence B
Started | 9 | 8
Completed | 9 | 7 (1 subject withdrew consent and left due to family emergencies)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sequence A: Period 1: Aminophylline 500 mg orally (corresponding to 395 mg theophylline), followed by 48 h washout period.
  Period 2: Ambrisentan 5 mg orally, followed by 48 h washout period.. Period 3: Aminophylline, 500 mg plus Ambrisentan, 5 mg orally, followed by 48 h washout period.
- Sequence B: Period 1: Ambrisentan 5 mg orally, followed by 48 h washout period. Period 2: Aminophylline 500 mg orally (corresponding to 395 mg theophylline), followed by 48 h washout period.
  Period 3: Aminophylline, 500 mg plus Ambrisentan, 5 mg orally, followed by 48 h washout period.
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Adverse Events Following Each Dose
Description: Dosing schedule:
  Aminophylline Alone (Single Dose of 500mg Aminophylline) Ambrisentan Alone (Single Dose of 5mg Ambrisentan) Ambrisentan and Aminophylline (Combined Single Dose of 500mg Aminophylline and 5mg Ambrisentan)
Time Frame: 48 h following each dose
Measure: Mean (Standard Deviation); unit: Mean number of adverse events
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 10 | 8
Mean number of adverse events
  Adverse Events after aminophylline | 2.5 (3.6) | 0.4 (0.7)
  Adverse Events after ambrisentan | 0.8 (1.3) | 0.4 (1.1)
  Adverse Events after combined treatment | 2.7 (3.7) | 0.5 (1.4)

2. Primary Outcome: Plasma Halflife of Theophylline (Aminophylline) and Ambrisentan When Administered Alone or in Combination
Description: Aminophylline Alone (Single Dose of 500mg Aminophylline) Aminophylline in Presence of Ambrisentan (Combined Single Dose of 500mg Aminophylline and 5mg Ambrisentan) Ambrisentan Alone (Single Dose of 5mg Ambrisentan) Ambrisentan in Presence of Aminophylline (Combined Single Dose of 500mg Aminophylline and 5mg Ambrisentan)
  Blood sample collections for plasma Ambrisentan and Theophylline determinations at 0-hour (pre-dose), and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Time Frame: 24 hours after dosing
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Aminophylline Alone | Aminophylline in Presence of Ambrisentan | Ambrisentan Alone | Ambrisentan in Presence of Aminophylline
Number analyzed (Participants) | 18 | 17 | 18 | 17
hours | 11.11 (3.15) | 9.96 (3.37) | 8.27 (1.72) | 9.12 (3.35)

3. Primary Outcome: Time Until Maximum Plasma Concentration (Tmax) of Theophylline (Aminophylline) and Ambrisentan When Administered Alone or in Combination
Description: as for outcome 2
Time Frame: 24h after dosing
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Aminophylline Alone | Aminophylline in Presence of Ambrisentan | Ambrisentan Alone | Ambrisentan in Presence of Aminophylline
Number analyzed (Participants) | 18 | 17 | 18 | 17
hours | 2.0 (0.8) | 1.50 (0.95) | 2.0 (1.09) | 2.0 (0.88)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Theophylline (Aminophylline) and Ambrisentan When Administered Alone or in Combination
Description: Aminophylline Alone (Single Dose of 500mg Aminophylline) Aminophylline in Presence of Ambrisentan (Combined Single Dose of 500mg Aminophylline and 5mg Ambrisentan) Ambrisentan Alone (Single Dose of 5mg Ambrisentan) Ambrisentan in Presence of Aminophylline (Combined Single Dose of 500mg Aminophylline and 5mg Ambrisentan)
Time Frame: 24h after dosing
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Aminophylline Alone | Aminophylline in Presence of Ambrisentan | Ambrisentan Alone | Ambrisentan in Presence of Aminophylline
Number analyzed (Participants) | 18 | 17 | 18 | 17
ng/ml | 6590 (1731.09) | 6780 (1519.16) | 464.5 (112.23) | 562 (110.90)

5. Primary Outcome: Area Under the Curve Within 24 Hours Post Dosing (AUC_0-24 Hours) of Theophylline (Aminophylline) and Ambrisentan When Administered Alone or in Combination
Description: as for outcome 2
Time Frame: 24h after dosing
Measure: Median (Standard Deviation); unit: h*ng/ml
Arm/Group | Aminophylline Alone | Aminophylline in Presence of Ambrisentan | Ambrisentan Alone | Ambrisentan in Presence of Aminophylline
Number analyzed (Participants) | 18 | 17 | 18 | 17
h*ng/ml | 75970.66 (16537.85) | 74451.38 (19726.55) | 3225.47 (700.84) | 3338.09 (837.03)

6. Primary Outcome: Area Under the Curve Post Dosing (AUC_0-infinity) of Theophylline (Aminophylline) and Ambrisentan When Administered Alone or in Combination
Description: as for outcome 2
Time Frame: 24h after dosing
Measure: Median (Standard Deviation); unit: h*ng/ml
Arm/Group | Aminophylline Alone | Aminophylline in Presence of Ambrisentan | Ambrisentan Alone | Ambrisentan in Presence of Aminophylline
Number analyzed (Participants) | 18 | 17 | 18 | 17
h*ng/ml | 99799.27 (28062.69) | 88545.08 (33678.29) | 3703.01 (866.21) | 3779.21 (977.93)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed starting from the time of first dosing, for the entire period of containment in the Duke Clinical Research Unit until discharge, and as part of the final visit.
Groups:
- Aminophylline Only: Aminophylline 500 mg orally (corresponding to 395 mg theophylline), followed by 48 h washout period.
- Ambrisentan Only: Ambrisentan 5 mg orally, followed by 48 h washout period. lowed by 48 h washout period.
- Combined Aminophylline and Ambrisentan: Combined single doses of Aminophylline 400 mg and ambrisentan 5 mg, followed by a 48 h washout period
Arm/Group | Aminophylline Only | Ambrisentan Only | Combined Aminophylline and Ambrisentan
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 5/18 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminophylline Only (N=18) | Ambrisentan Only (N=18) | Combined Aminophylline and Ambrisentan (N=18)
Cramping (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (3) | 2 (5)
Headache (Nervous system disorders) | 2 (2) | 5 (6) | 2 (3)
Tremors (Nervous system disorders) | 4 (7) | 0 (0) | 2 (3)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4)
Dizziness/ lightheadedness (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Palpitations and Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Facial flushing and hot flashes (General disorders) | 0 (0) | 1 (1) | 1 (2)
Sweaty clammy hands and feet (General disorders) | 0 (0) | 0 (0) | 2 (3)
Feeling different and increased energy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety and restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hiccups (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Liver safety panel (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) — Total bilirubin, AST (serum aspartate transaminase), and ALT (alanine transaminase) were investigated within 48 hours of dosing for elevation to more than 3 x the upper limit of normal range.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No